CLINICAL TRIAL: NCT03243123
Title: Passive Mobilization With Robotic Assistance Improve Hemiparetic Upper Limb Circulation and Functional Status in Stroke Survivors.
Brief Title: Upper Limb Robotic Rehabilitation After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, Massimiliano Gobbo, MD, Università degli Studi di Brescia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201701
Record Dates: First submitted 2017-08-03; First posted 2017-08-08 (Actual); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Passive mobilization (Experimental): Upper limb passive mobilization assisted with robotic device
  Interventions: Device: Robotic passive mobilization

INTERVENTIONS:
Device: Robotic passive mobilization — The intervention was performed using the Gloreha (Idrogenet, Italy) robotic system. The system consists of a soft exoskeleton similar to a glove. Passive hand joints mobilization is provided by a hydraulic system. Each patient underwent a session of 20 min passive mobilization of the paretic hand.

SUMMARY:
This is a single arm study aimed at evaluating the acute effects induced by a single session of robot-assisted passive hand mobilization on local perfusion and upper limb function in post-stroke hemiparetic patients. Twenty-three participants with subacute or chronic stroke received 20 min passive mobilization of the paretic hand with robotic assistance. After the intervention, significant improvements were found in forearm perfusion, muscle tone significantly decreased and subjects reported decreased upper limb heaviness, stiffness and pain. This study supports novel evidence that hand robotic assistance promotes local forearm circulation, may help in the management of spasticity and acutely alleviates reported symptoms of heaviness, stiffness and pain in subjects with post-stroke hemiparesis.

ELIGIBILITY:
Inclusion Criteria:

* first event of cerebrovascular stroke; unilateral paresis; ability to remain in sitting position

Exclusion Criteria:

* bilateral impairment; cognitive or behaviorql dysfunctions; finger flexion contracture; degenerative or non degenerative neurological conditions; refusal or inability to provide informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2014-11-15 (Actual); Study Completion 2014-12-23 (Actual)

PRIMARY OUTCOMES:
Forearm perfusion | 30 minutes
  Amount of total hemoglobin circulating in the forearm muscle tissues.
Muscle tone | 30 minutes
  The tone of the muscle assessed with Modified Ashworth Scale

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gobbo M, Gaffurini P, Vacchi L, Lazzarini S, Villafane J, Orizio C, Negrini S, Bissolotti L. Hand Passive Mobilization Performed with Robotic Assistance: Acute Effects on Upper Limb Perfusion and Spasticity in Stroke Survivors. Biomed Res Int. 2017;2017:2796815. doi: 10.1155/2017/2796815. Epub 2017 Sep 28. PMID 29094043